CLINICAL TRIAL: NCT02784145
Title: Effects of Resistant Starch on Bowel Habits, Fecal Short Chain Fatty Acids and Gut Microbiota in Parkinson Disease
Acronym: RESISTA-PD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universität des Saarlandes (Other)
Responsible Party: Principal Investigator, Dr. Marcus Unger, PD Dr., Universität des Saarlandes
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RESISTA-PD
Record Dates: First submitted 2016-05-17; First posted 2016-05-26 (Estimated); Last update posted 2018-05-15 (Actual); Status verified 2018-05

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Resistant Starch

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- RS (Other): Resistant starch supplementation (5 g twice a day)
  Interventions: Dietary Supplement: Resistant starch
- No RS (Other): PD patients who do not receive resistant starch, but who receive recommendations concerning healthy Nutrition (based on the guidelines of the German Society for Nutrition)
  Interventions: Other: Recommendation with regard to nutrition

INTERVENTIONS:
Dietary Supplement: Resistant starch
  Arms: RS
Other: Recommendation with regard to nutrition — Subjects in this arm will receive General recommendations with regard to nutrition based on the guidlines of the German Society for nutrition
  Arms: No RS

SUMMARY:
The investigators will investigate the effects of an 8-week resistant starch (RS) supplementation (5 g twice a day) in patients with Parkinson Disease and matched controls on:

1. symptoms of constipation (assessed by clinical scores);
2. fecal short chain fatty acid concentrations (measured by chromatography);
3. gut microbiota composition.

ELIGIBILITY:
Main Inclusion Criteria:

* Written informed to participate
* For patients: diagnosis of Parkinson Disease

Main Exclusion Criteria:

* Use of antibiotics, steroids or probiotic supplements
* Chronic or acute disorders of the gastrointestinal tract
* History of gastrointestinal surgery (other than appendectomy)
* For healthy controls: Family history of neurodegenerative disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2016-05; Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Bowel habits | 8 weeks
  Number of patients with improved bowel habits
Fecal short chain fatty acid (SCFA) concentrations | 8 weeks
  Number of patients with either a) increased, b.) unaltered or c) decreased concentration of short chain fatty acids in fecal samples at 8 weeks (compared to baseline)
Analysis of fecal microbiota composition | 8 weeks
  Analysis to detect changes between baseline and 8 weeks of resistant starch supplementation

CONTACTS AND LOCATIONS:
Overall Officials: Marcus M Unger, PD Dr. med., Principal Investigator — Saarladnd University, Department of Neurology
Locations (1):
- Saarland University, Homburg / Saar, Saarland, Germany

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Becker A, Schmartz GP, Groger L, Grammes N, Galata V, Philippeit H, Weiland J, Ludwig N, Meese E, Tierling S, Walter J, Schwiertz A, Spiegel J, Wagenpfeil G, Fassbender K, Keller A, Unger MM. Effects of Resistant Starch on Symptoms, Fecal Markers, and Gut Microbiota in Parkinson's Disease - The RESISTA-PD Trial. Genomics Proteomics Bioinformatics. 2022 Apr;20(2):274-287. doi: 10.1016/j.gpb.2021.08.009. Epub 2021 Nov 25. PMID 34839011